CLINICAL TRIAL: NCT05410834
Title: The Characterization of Pro-vascular Regenerative Cell Exhaustion in Women With Polycystic Ovarian Syndrome
Brief Title: Pro-vascular Regenerative Cell Exhaustion in Women With Polycystic Ovarian Syndrome
Acronym: PCOS-RCE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00063366
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovarian syndrome; Progenitor cells; Women's Health; Insulin resistance; Chronic disease
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Chronic Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples to be retained for 5 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with polycystic ovarian syndrome: Individuals with a documented diagnosis of polycystic ovarian syndrome
- Individuals without polycystic ovarian syndrome: Individuals without a known diagnosis of polycystic ovarian syndrome but with regular menstrual cycles

SUMMARY:
PCOS-RCE is an observational, cross-sectional, two-arm study that is aimed at determining if an established diagnosis of polycystic ovarian syndrome (PCOS) influences the number of blood vessel-forming stem cells in the bloodstream. Circulating progenitor cells will be enumerated and the distribution patterns of these cell types will be assessed to determine if these parameters differ between individuals with PCOS and individuals without PCOS. Specifically, this study will evaluate if differential regenerative cell exhaustion (RCE) may account, at least in part, for the differences in cardiovascular risk reported between individuals with a diagnosis of PCOS and those without.

DETAILED DESCRIPTION:
Individuals with polycystic ovarian syndrome (PCOS) have been reported to be at higher risk of cardiovascular disease when compared to those without PCOS. While differential environmental exposures and genetic morphometries are believed to account in part for the difference, there is growing evidence that cardiometabolic risk factors can accelerate pro-vascular progenitor cell depletion and dysfunction. The cumulative effects that aberrant regenerative cell exhaustion (RCE) have on vessel repair accordingly increases the risk of atherothrombotic events.

PCOS-RCE is an observational, cross-sectional, two-arm study that will evaluate the progenitor cell profiles of peripheral blood samples from 30 individuals (15 with PCOS, 15 without PCOS). The working hypothesis is that individuals with PCOS have innately different progenitor cell profiles that can be further altered by their environment and genotype. The resultant differences in RCE capability will affect the balance between pro-inflammatory and vessel repair functions that, in turn, contribute to the contrasting cardiometabolic risks exhibited between the two study cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to provide informed consent
* Females aged 30 and above
* Must meet criteria for one of the following two groups:

  1. Documented diagnosis of PCOS OR
  2. Normal and regular menstrual cycles with no known diagnosis of PCOS

Exclusion Criteria:

* Menopause, as defined by 12 months of amenorrhea
* Known causes of irregular menstrual bleeding caused by conditions other than PCOS
* Known secondary causes of ovulatory dysfunction and/or hyperandrogenism
* Current pregnancy, active lactation, or less than 6 months postpartum
* Ongoing treatment with ovulation-inducing medication
* History of hysterectomy and/or bilateral oophorectomy
* Severe congestive heart failure (as defined by New York Heart Association - class IV)
* Any life-threatening disease expected to result in death within the next 2 years
* Any malignancy not considered cured. A subject is considered cured if there has been no evidence of cancer recurrence for the 5 years prior to screening.
* Known severe liver disease
* Known acquired immunodeficiency syndrome such as HIV
* Current treatment with systemic or oral corticosteroid therapy or other immunosuppressive agents
* Known autoimmune disorder (exception: type 1 diabetes)
* Active infectious disease requiring antibiotic or anti-viral agents

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from primary care clinics in the Greater Toronto Area using paper-based and electronic medical records.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of circulating ALDHhiSSChi granulocytes | Baseline
  Difference in the frequency of circulating ALDHhi SSChi granulocytes between women with PCOS versus without PCOS

SECONDARY OUTCOMES:
Number of circulating ALDHhiSSCmid monocytes | Baseline
  Difference in the number of circulating ALDHhi SSCmid monocytes with M1 vs M2 polarization between women with PCOS versus without PCOS
Number of circulating ALDHhiSSClo primitive progenitor cells | Baseline
  Difference in the number of circulating ALDHhi SSClo primitive progenitor cells in women with PCOS versus without PCOS

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD, PhD, Principal Investigator — University of Toronto; David A Hess, PhD, Principal Investigator — University of Western Ontario, Canada
Locations (3):
- Canada (3):
  - Centrum Services Newmarket, Newmarket, Ontario
  - Diagnostic Assessment Centre, Scarborough Village, Ontario
  - Langstaff Medical Centre, Woodbridge, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vassalli G. Aldehyde Dehydrogenases: Not Just Markers, but Functional Regulators of Stem Cells. Stem Cells Int. 2019 Jan 13;2019:3904645. doi: 10.1155/2019/3904645. eCollection 2019. PMID 30733805
- [Background] Bajuk Studen K, Pfeifer M. Cardiometabolic risk in polycystic ovary syndrome. Endocr Connect. 2018 Jul;7(7):R238-R251. doi: 10.1530/EC-18-0129. Epub 2018 May 29. PMID 29844207
- [Background] Rudnicka E, Suchta K, Grymowicz M, Calik-Ksepka A, Smolarczyk K, Duszewska AM, Smolarczyk R, Meczekalski B. Chronic Low Grade Inflammation in Pathogenesis of PCOS. Int J Mol Sci. 2021 Apr 6;22(7):3789. doi: 10.3390/ijms22073789. PMID 33917519
- [Background] Murri M, Luque-Ramirez M, Insenser M, Ojeda-Ojeda M, Escobar-Morreale HF. Circulating markers of oxidative stress and polycystic ovary syndrome (PCOS): a systematic review and meta-analysis. Hum Reprod Update. 2013 May-Jun;19(3):268-88. doi: 10.1093/humupd/dms059. Epub 2013 Jan 9. PMID 23303572
- [Background] Terenzi DC, Al-Omran M, Quan A, Teoh H, Verma S, Hess DA. Circulating Pro-Vascular Progenitor Cell Depletion During Type 2 Diabetes: Translational Insights Into the Prevention of Ischemic Complications in Diabetes. JACC Basic Transl Sci. 2018 Nov 5;4(1):98-112. doi: 10.1016/j.jacbts.2018.10.005. eCollection 2019 Feb. PMID 30847424
- [Background] Balber AE. Concise review: aldehyde dehydrogenase bright stem and progenitor cell populations from normal tissues: characteristics, activities, and emerging uses in regenerative medicine. Stem Cells. 2011 Apr;29(4):570-5. doi: 10.1002/stem.613. PMID 21308868
- [Background] Qadura M, Terenzi DC, Verma S, Al-Omran M, Hess DA. Concise Review: Cell Therapy for Critical Limb Ischemia: An Integrated Review of Preclinical and Clinical Studies. Stem Cells. 2018 Feb;36(2):161-171. doi: 10.1002/stem.2751. Epub 2018 Jan 3. PMID 29226477
- [Background] Putman DM, Cooper TT, Sherman SE, Seneviratne AK, Hewitt M, Bell GI, Hess DA. Expansion of Umbilical Cord Blood Aldehyde Dehydrogenase Expressing Cells Generates Myeloid Progenitor Cells that Stimulate Limb Revascularization. Stem Cells Transl Med. 2017 Jul;6(7):1607-1619. doi: 10.1002/sctm.16-0472. Epub 2017 Jun 15. PMID 28618138
- [Background] Terenzi DC, Bakbak E, Trac JZ, Al-Omran M, Quan A, Teoh H, Verma S, Hess DA. Isolation and characterization of circulating pro-vascular progenitor cell subsets from human whole blood samples. STAR Protoc. 2021 Feb 1;2(1):100311. doi: 10.1016/j.xpro.2021.100311. eCollection 2021 Mar 19. PMID 33554145
- [Background] Xiong YL, Liang XY, Yang X, Li Y, Wei LN. Low-grade chronic inflammation in the peripheral blood and ovaries of women with polycystic ovarian syndrome. Eur J Obstet Gynecol Reprod Biol. 2011 Nov;159(1):148-50. doi: 10.1016/j.ejogrb.2011.07.012. Epub 2011 Sep 9. PMID 21908093
- [Background] Mohammadi M. Oxidative Stress and Polycystic Ovary Syndrome: A Brief Review. Int J Prev Med. 2019 May 17;10:86. doi: 10.4103/ijpvm.IJPVM_576_17. eCollection 2019. PMID 31198521
- [Background] Capoccia BJ, Robson DL, Levac KD, Maxwell DJ, Hohm SA, Neelamkavil MJ, Bell GI, Xenocostas A, Link DC, Piwnica-Worms D, Nolta JA, Hess DA. Revascularization of ischemic limbs after transplantation of human bone marrow cells with high aldehyde dehydrogenase activity. Blood. 2009 May 21;113(21):5340-51. doi: 10.1182/blood-2008-04-154567. Epub 2009 Mar 26. PMID 19324906
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Background] Hess DA, Wirthlin L, Craft TP, Herrbrich PE, Hohm SA, Lahey R, Eades WC, Creer MH, Nolta JA. Selection based on CD133 and high aldehyde dehydrogenase activity isolates long-term reconstituting human hematopoietic stem cells. Blood. 2006 Mar 1;107(5):2162-9. doi: 10.1182/blood-2005-06-2284. Epub 2005 Nov 3. PMID 16269619
- [Background] Hess DA, Terenzi DC, Trac JZ, Quan A, Mason T, Al-Omran M, Bhatt DL, Dhingra N, Rotstein OD, Leiter LA, Zinman B, Sabongui S, Yan AT, Teoh H, Mazer CD, Connelly KA, Verma S. SGLT2 Inhibition with Empagliflozin Increases Circulating Provascular Progenitor Cells in People with Type 2 Diabetes Mellitus. Cell Metab. 2019 Oct 1;30(4):609-613. doi: 10.1016/j.cmet.2019.08.015. Epub 2019 Aug 30. PMID 31477497
- [Background] Aboeldalyl S, James C, Seyam E, Ibrahim EM, Shawki HE, Amer S. The Role of Chronic Inflammation in Polycystic Ovarian Syndrome-A Systematic Review and Meta-Analysis. Int J Mol Sci. 2021 Mar 8;22(5):2734. doi: 10.3390/ijms22052734. PMID 33800490
- [Background] Putman DM, Liu KY, Broughton HC, Bell GI, Hess DA. Umbilical cord blood-derived aldehyde dehydrogenase-expressing progenitor cells promote recovery from acute ischemic injury. Stem Cells. 2012 Oct;30(10):2248-60. doi: 10.1002/stem.1206. PMID 22899443
- [Background] Terenzi DC, Trac JZ, Teoh H, Gerstein HC, Bhatt DL, Al-Omran M, Verma S, Hess DA. Vascular Regenerative Cell Exhaustion in Diabetes: Translational Opportunities to Mitigate Cardiometabolic Risk. Trends Mol Med. 2019 Jul;25(7):640-655. doi: 10.1016/j.molmed.2019.03.006. Epub 2019 Apr 30. PMID 31053416